CLINICAL TRIAL: NCT00633204
Title: Phase II Study of Bladder Cancer Using Novel Tumor Antigens for Prevention of the Recurrence for Bladder Cancer After TUR-Bt
Brief Title: Peptide Vaccine Focusing on Prevention of the Recurrence for Bladder Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Iwate Medical University (Other)
Collaborators: Human Genome Center, Institute of Medical Science, University of Tokyo (Other)
Responsible Party: Department of Urology, Iwate Medical University
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: IMU-H18-59-P2
Record Dates: First submitted 2008-03-04; First posted 2008-03-11 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2009-01

CONDITIONS: Bladder Cancer
Keywords: Epitope peptide, CTL, TUR-Bt, Bladder cancer, Vaccination; Bladder cancer after surgery
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — KIF20B protein, human; DEPDC1 protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: MPHOSPH1 and DEPDC1 — DEPDC1-9-294, and/or MPHOSPH1-9-278 will be administered by subcutaneously injection once every week after curative surgery 8 times and BCG in bladder simultaneously. Then, DEPDC1-9-294, and/or MPHOSPH1-9-278 will be administered once every month. These peptides are determined to administer in accordance with the protein expression using immunohistochemical staining. These peptides are conjugated with Montanide ISA 51 as an adjuvant.

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy for the prevention of the recurrence for bladder cancer after TUR-Bt

DETAILED DESCRIPTION:
DEP domain containing 1(DEPDC1) and M phase phosphoprotein 1(MPHOSPH1) have been identified using genome-wide expression profile analysis by the use of cDNA microarray in our previous studies. The investigators have determined the HLA-A*2402 restricted epitope peptides derived from DEPDC1, DEPDC1-9-294, and MPHOSPH1, MPHOSPH1-9-278. These epitopes showed strong IFN-g production when stimulated with the appropriate targets expressed the appropriate protein and HLA-A*2402. Furthermore, when vaccinated these peptides, specific CTLs were determined after the vaccination. Therefore we focused on the prevention of the recurrence of the bladder cancer after surgery using these peptides.

ELIGIBILITY:
Inclusion Criteria DISEASE CHARACTERISTICS

1. Bladder cancer without solitary and low grade tumor
2. Protein expression of MPHOSPH1 and DEPDC1 on the tumor

PATIENTS CHARACTERISTICS

1. Patients must be treated completely by Transurethral resection of the bladder tumor(TUR-Bt), and must have no residual tumor after re-TUR-Bt.
2. Patients without the first time, solitary, low grade1 bladder cancer, which tumor is diagnosed histologically transitional cell carcinoma of bladder.
3. Patients must be treated by TUR-BT, who are able to treated by Intravesical Bacillus calmette-guerin (BCG) for adjuvant therapy
4. ECOG performance status of 0 to 1
5. Age ≥ 20 years, ≤80 years
6. WBC≥ 2,000/mm³, ≤15000/mm³ Platelet count ≥ 75000/mm³ AST, ALT ≤150 IU/l Total bilirubin ≤ 3.0 mg/dl Creatinine ≤ 3.0 mg/dl
7. Samples of bladder cancer must express MPHOSPH1 or DEPDC1
8. Able and willing to give valid written informed consent

Exclusion Criteria:

1. Pregnancy (women of childbearing potential: Refusal or inability to use effective means of contraception)
2. Breastfeeding
3. Patients willing to childbearing ( Refusal or inability to use effective means of contraception)
4. Serious infections requiring antibiotics
5. Concomitant treatment with steroids or immunosuppressing agent
6. Other malignancy difficult to control.
7. Decision of unsuitableness by principal investigator or physician-in-charge

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-02; Primary Completion 2011-11 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate after surgery (TUR-BT) | 2 years

SECONDARY OUTCOMES:
feasibility | 2 years
CTL response | 2 years
CD8 population | 2 years
Change in level of regulatory T cells | 2 years
Overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Tomoaki Fujioka, M.D. & Ph.D., Study Chair — Department of Urology, Iwate Medical University
Locations (1):
- Iwate Medical University School of Medicine, Morioka, Iwate, Japan

REFERENCES:
- [Result] Kanehira M, Katagiri T, Shimo A, Takata R, Shuin T, Miki T, Fujioka T, Nakamura Y. Oncogenic role of MPHOSPH1, a cancer-testis antigen specific to human bladder cancer. Cancer Res. 2007 Apr 1;67(7):3276-85. doi: 10.1158/0008-5472.CAN-06-3748. PMID 17409436
- [Result] Kanehira M, Harada Y, Takata R, Shuin T, Miki T, Fujioka T, Nakamura Y, Katagiri T. Involvement of upregulation of DEPDC1 (DEP domain containing 1) in bladder carcinogenesis. Oncogene. 2007 Sep 27;26(44):6448-55. doi: 10.1038/sj.onc.1210466. Epub 2007 Apr 23. PMID 17452976